CLINICAL TRIAL: NCT03799835
Title: An Open Label, Randomized, Phase III Trial, Evaluating Efficacy of Atezolizumab in Addition to One Year BCG (Bacillus CaLmette-Guerin) Bladder Instillation in BCG-naive Patients With High-risk Non-muscle Invasive Bladder cANcer
Brief Title: Atezolizumab Plus One-year BCG Bladder Instillation in BCG-naive High-risk Non-muscle Invasive Bladder Cancer Patients
Acronym: ALBAN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1717; 2017-004512-19 (EudraCT Number)
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A : control arm (Active Comparator): BCG therapy only
  BCG therapy will be administered in two phases:
  * induction phase: weekly administration of full dose of BCG intravesically up to 6 weeks, starting on the day of the first induction instillation (D1)
  * maintenance phase: full-dose BCG administered once per week for 3 weeks, at week 13 (i.e. 3 months after the first BCG instillation of induction, D1), at week 26 (6 months from D1) and week 52 (12 months from D1).
  Interventions: Drug: BCG
- Arm B: experimental arm (Experimental): BCG therapy + administration of atezolizumab
  1. BCG therapy will be administered in two phases:
     * induction phase: weekly administration of full dose of BCG intravesically up to 6 weeks, starting on the day of the first induction instillation (D1)
     * maintenance phase: full-dose BCG administered once per week for 3 weeks, at week 13 (i.e. 3 months after the first BCG instillation of induction, D1), at week 26 (6 months from D1) and week 52 (12 months from D1).
  2. atezolizumab is administered by IV infusion every 3 weeks (21 [± 2] days) for 1 year (18 cycles as a maximum).
  Interventions: Drug: BCG; Drug: Atezolizumab

INTERVENTIONS:
Drug: BCG — Intravesical administration OncoTice wil be used only under two conditions : BCG Medac® unavailable and the patient has received at minimum one instillation of BCG Medac®
  Other Names: Bacillus Calmette Guerin (BCG) Medac®; OncoTice
Drug: Atezolizumab — IV perfusion
  Other Names: MPDL3280A; Tecentriq®
  Arms: Arm B: experimental arm

SUMMARY:
This is an open-label, randomized, multicentric study in patients with high-risk non-muscle invasive bladder cancer who had never received BCG for this disease.

The primary objective is to evaluate the efficacy of atezolizumab as measured by Event-Free survival.

DETAILED DESCRIPTION:
ALBAN study recruited 517 patients in 45 centers in Europe (France, Belgium and Spain), according to a ratio 1:1 in the following arms of treatment:

* Arm A (control arm): BCG only
* Arm B (experimental arm): BCG+ atezolizumab

The are two factors of stratifications (center and CIS).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form after the last endoscopic surgery (TURBT)
2. Adult man and women ( age ≥18 years)
3. Any high risk non muscle invasive urothelial carcinoma histologically confirmed (mixed histology tumors allowed if urothelial carcinoma histology is predominant) defined on the TURBT as any of the following :

   * T1 tumor and/or
   * High grade (WHO 2004) and/or
   * Grade 3 (WHO1973) and/or
   * Carcinoma in situ (CIS)
4. Tumor tissue available from the surgery for central confirmation of the diagnosis and analysis the expression of PD-L1
5. At least one additional (second) resection of the primary tumor has been performed in any of the following cases [without upstaging towards Muscle Invasive Bladder Cancer (EAU guidelines, 2017)] :

   * T1 tumors at physician's discretion,
   * incomplete initial TURB,
   * no muscle in the specimen (can be omitted if TaLG/G1 tumors or primary CIS only was found)
6. Absence of metastasis in pelvis, abdomen, or chest, as confirmed by a negative baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan no more than 90 days prior to the first study treatment
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
8. Life expectancy ≥12 weeks
9. Systolic blood pressure (BP) <160 mmHg and diastolic BP <95 mmHg, as documented within 7 days prior to the first study treatment (hypertension allowed provided it is controlled)
10. Adequate hematologic and end-organ function, as defined by the following laboratory results obtained within 7 days prior to the first study treatment:

    * absolute neutrophil count (ANC) ≥1500 cells/μL
    * white blood cell (WBC) counts >2500/μL
    * Lymphocyte count ≥300/μL
    * Platelet count ≥100,000/μL
    * Hemoglobin ≥9.0 g/dL
    * aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), and alkaline phosphatase ≤2.5 × the upper limit of normal (ULN)
    * Serum bilirubin ≤1.0 × ULN Patients with known Gilbert disease who have serum bilirubin level ≤3 × ULN may be enrolled.
    * Partial thromboplastin time (PTT)/Prothrombin Time (PT) ≤1.5 × ULN or international normalized ratio (INR) <1.7 × ULN
    * Calculated creatinine clearance ≥20 mL/min (Cockcroft-Gault formula)
11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab
12. Patients affiliated to the social security system
13. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

1. Patient having received previous BCG therapy for bladder cancer
2. Any approved anti-cancer therapy, including systemic chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment. Hormone-replacement therapy or oral contraceptives are allowed
3. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or five half-lives of the drug, whichever is longer, prior to day 1 of study treatment
4. Malignancies other than urothelial cancer within 5 years prior to Day 1 of cycle 1 of treatment except the following:

   * Patients with localized low risk prostate cancer (defined as Stage ≤T2b, Gleason score ≤7, and PSA at prostate cancer diagnosis ≤20 ng/mL [if measured]) treated with curative intent (radiotherapy and/or prostatectomy) and without prostate-specific antigen (PSA) recurrence are eligible.
   * Patients with low risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤7 and PSA ≤10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
   * Patients with malignancies of a negligible risk of metastasis or death (e.g., risk of metastasis or death <5% at 5 years) are eligible provided they meet all of the following criteria: malignancy treated with expected curative intent (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) and no evidence of recurrence or metastasis by follow-up imaging and any disease-specific tumor markers.
5. Pregnancy or breastfeeding
6. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
7. Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
8. History of autoimmune disease or history of immunosuppression, or conditions associated with congenital or acquired immune deficiency , including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (see Appendix 6 for a more comprehensive list of autoimmune diseases)

   * Patients with a history of autoimmune-related hypothyroidism/hyperthyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
   * Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
   * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan may be eligible.
   * History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
9. Serum albumin <2.5 g/dL
10. Known HIV infection
11. Patients with active hepatitis B virus (HBV; chronic or acute; defined as having a positive hepatitis B surface antigen (HBsAg) test prior the randomisation) or hepatitis C.

    * Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody (HBc Ab) and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to randomisation.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
12. Known active tuberculosis
13. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
14. Signs or symptoms of urinary infection and/or other signs and symptoms > grade 1 (NCI CTCAE v5.0) within 2 weeks prior to Cycle 1, Day 1

    * Patients receiving therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1 are not eligible
    * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
15. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months before Cycle1, Day 1, unstable arrhythmias, or unstable angina.

    - Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
16. Major surgical procedure other than for diagnosis within 4 weeks prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
17. Prior allogeneic stem cell or solid organ transplant
18. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation if such a live, attenuated vaccine will be required during the study

    - Influenza vaccination should be given during influenza season only (approximately October through May in the Northern Hemisphere and approximately April through September in the Southern Hemisphere). Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1, at randomization, during treatment or within 5 months following the last dose of atezolizumab (for patients randomized to atezolizumab).
19. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
20. Prior treatment with CD137 agonists or immune checkpoint-blockade therapies, including anti-CD40, anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
21. Treatment with systemic immunostimulatory agents (including but not limited to interferons, interleukin 2 (IL-2)) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1
22. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial

    * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea, multiple doses for contrast allergy) may be enrolled in the study.
    * The use of inhaled or low-dose (e.g., ≤10 mg/day prednisone) corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, mineralocorticoids (e.g., fludrocortisone for adrenal insufficiency) and low-dose corticosteroids for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
23. Person deprived of their liberty or under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival | 5 years
  The primary efficacy endpoint is event-free survival defined as the time from randomization to the time of first event-free survival (EFS) event restricted to high grade or low grade Ta tumor at any time after the start of therapy; T1 tumor and higher (e.g .T2) at any time after the start of therapy; CIS tumor at least 6 months after the start of therapy ( Persistent CIS without papillary tumor at 3 months without any other event for EFS will not be an event); any UTUC after NMIBC; any N+ at any time after the start of therapy; any M+ at any time after the start of therapy; or death whatever the cause.

SECONDARY OUTCOMES:
High-grade recurrence-free survival | 5 years
  High-grade recurrence-free survival is defined by reappearance of high-grade risk disease (high grade, T1 or CIS) or death.
Progression-free survival | From randomization to the date of progression, assessed up to 5 years
  Progression- free survival defined as the time from randomization to the date of disease progression defined as increase of stage from Ta to T1 or from CIS to T1; progression to Muscle Invasive Bladder Cancer (T≥ 2) or to lymph node N+ or to distant disease M+; the date of progression being determined by the endoscopic resection (TURBT) for a local relapse or by CT scan in case of non-local relapse.
Disease-specific survival | From randomization to the date of death, assessed up to 5 years
  Disease-specific survival defined as the time from randomization to the date of death from bladder cancer.
Overall Survival | From randomization to the date of death, assessed up to 5 years
  Overall Survival defined as the time from randomization to the date of death from any cause.
Disease worsening in each arm | From randomization to the date of death, assessed up to 5 years
  Disease worsening, defined as cystectomy or change in therapy indicative, including systemic chemotherapy or radiation therapy. The date of diagnosis (cystoscopy or CT scan) leading to cystectomy or chemotherapy will be considered as the time of disease worsening.
Complete response in each arm | 6 weeks and 2 years after randomization
  Complete response is assessed by cystoscopy and cytology.
Complete response among patients with CIS | 6 weeks and 2 years after randomization
  Complete response is assessed by cystoscopy and cytology.
National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | Throughout study completion, assessed up to 5 years
  The frequency, nature, and severity of adverse events graded according to NCI CTCAE v5.0 and according to the immune-related adverse event (irAE).
Quality of life questionnaire (QLQ): QLQ-C30 questionnaire (EORTC) | At randomization, every 12 weeks for years 1 and 2 after randomization, then every 24 weeks for years 3 to 5 after randomization
  This self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Roupret, MD-PHD, Principal Investigator — Hôpital Pitié-Salpétrière; Yohann Loriot, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (38):
- Belgium (2):
  - Groupe Jolimont - Hôpital de Jolimont, Haine-Saint-Paul
  - AZ Delta - Campus Rumbeke, Roeselare
- France (30):
  - Centre Hospitalier Universitaire Angers, Angers
  - Centre Hospitalier Universitaire Bordeaux, Bordeaux
  - Hôpital G. Montpied, Clermont-Ferrand
  - Clinique Claude Bernard, Ermont
  - CHU Grenoble, Grenoble
  - Hôpital privé Toulon - Sainte Marguerite, Hyères
  - Hôpital du Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint Vincent, Lille
  - Hôpital privé de la Louvière, Lille
  - Hôpital Saint Philibert, Lomme
  - Insitut Paoli Calmette, Marseille
  - Centre Hospitalier Universitaire Marseille, Marseille
  - Centre Hospitalier Universitaire Nîmes, Nîmes
  - Hôpital européen Georges Pompidou, Paris
  - Hôpital Saint Louis, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hôpital Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Universitaire Tenon, Paris
  - Hôpital Diaconesses- Croix Saint Simon, Paris
  - Hôpital La Pitié Salpétrière, Paris
  - Centre Hospitalier Universitaire Lyon Sud, Pierre-Bénite
  - Centre CARIO-HPCA, Plérin
  - Centre Hospitalier Universitaire Rennes, Rennes
  - Hôpitaux d'instruction des armées Begin, Saint-Mandé
  - Hôpital Foch, Suresnes
  - Hôpitaux Leman, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Spain (6):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Jerez de la Frontera, Cadiz
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients